CLINICAL TRIAL: NCT06674785
Title: Effects of Extracorporeal Shock Wave Therapy on Shoulder Internal Rotator Spasticity in Post-Stroke Patients: A Randomized Controlled Trial
Brief Title: SIRS-ESWT Trial: Shoulder Internal Rotator Spasticity Trial Treated With Extracorporeal Shock Wave Therapy Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202409035RIND
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-10

CONDITIONS: Stroke; Muscle Spasticity
Keywords: stroke; spasticity; shock wave; shoulder
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant Care Provider Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Focused Extracorporeal Shock Wave (Experimental): Participants in this arm will receive focused Extracorporeal Shock Wave Therapy (ESWT) targeting four specific muscles: subscapularis, pectoralis major, latissimus dorsi, and teres major muscles. Each muscle will receive 1,000 shockwave shots per session, accumulating to a total of 4,000 shots across all targeted muscles in each session. The treatment will be administered twice a week for two consecutive weeks, resulting in a total of four treatment sessions.
  Interventions: Device: focused extracorporeal shock wave therapy (ESWT)
- Placebo-Controlled Shockwave Therapy (Placebo Comparator): Participants in this arm will receive placebo-controlled focused ESWT, mirroring the treatment protocol of the experimental group but without the application of active shockwaves.
  Interventions: Device: focused extracorporeal shock wave therapy (ESWT)

INTERVENTIONS:
Device: focused extracorporeal shock wave therapy (ESWT) — The focused shockwaves are directed at the affected muscles in the upper limb, specifically targeting the subscapularis, pectoralis major, latissimus dorsi, and teres major muscles.
  Arms: Focused Extracorporeal Shock Wave
Device: focused extracorporeal shock wave therapy (ESWT) — Placebo shockwave therapy directed at subscapularis, pectoralis major, latissimus dorsi, and teres major muscles.
  Arms: Placebo-Controlled Shockwave Therapy

SUMMARY:
Extracorporeal shock wave therapy (ESWT) has shown potential in reducing post-stroke limb spasticity. This study aims to evaluate the efficacy of focused ESWT on shoulder internal rotator spasticity in post-stroke patients.

DETAILED DESCRIPTION:
This study aimed to evaluate the effects of focused extracorporeal shock wave therapy (ESWT) on shoulder internal rotator spasticity in stroke patients. Participants were randomized into two groups: an experimental group receiving targeted ESWT on specific shoulder internal rotators, and a control group receiving placebo treatments mimicking the shockwave therapy, with treatments administered twice weekly over two weeks for a total of four sessions.

The efficacy of the treatment was measured using a comprehensive set of assessment tools, including range of motion, pain levels, spasticity scales, functional assessments, as well as measures of daily living activities, and ultrasound strain elastography. The outcomes were evaluated at multiple points in time: before treatment, and 1, 4, 12, and 24 weeks after the therapy concluded, to assess both immediate and sustained effects of the treatment on shoulder function and spasticity in stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with unilateral cerebral stroke.
* Restricted passive external rotation of the spastic shoulder by more than 20 degrees.
* A Modified Ashworth Scale score of 1 or higher for shoulder internal rotator spasticity.
* Stable medical condition and vital signs.
* Clear consciousness, able to follow instructions.

Exclusion Criteria:

* History of two or more strokes, traumatic brain injury, brain tumors, or other cerebral disorders.
* Coexisting central nervous system disorders (e.g., spinal cord injury, Parkinson's disease) or other musculoskeletal conditions affecting muscle tone assessment.
* Ineligibility for shock wave intervention due to malignancies, coagulation disorders, localized infections, or presence of a pacemaker.
* Prior shock wave intervention or botulinum toxin injection for post-stroke spasticity within the past three months.
* Inability to participate in interventions or functional assessments due to cognitive, consciousness, or language impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
passive range of motion for the shoulder joints | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  the extent to which a joint can be moved without the patient actively participating in the movement
shoulder strength | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  the muscle power generated by the shoulder muscles, quantified using the Medical Research Council (MRC) scale, which grades muscle strength from 0 (no visible contraction) to 5 (normal strength against full resistance)
Visual Analogue Scale (VAS) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  individuals rate their pain from 0 to 10, where 0 represents 'no pain' and 10 signifies 'the worst pain imaginable
modified Ashworth scale (MAS) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  Evaluate spasticity in individuals with neurological conditions. The scale ranges from 0, indicating no increase in muscle tone, to 4, which represents severe spasticity with affected parts rigid in flexion or extension.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment for the Upper Extremity (FMA-UE) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  range from 0 (complete paralysis) to 66 (full function), assessing motor recovery in post-stroke upper extremities
Action Research Arm Test (ARAT) | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  a standardized measure evaluating upper limb motor ability in stroke patients, scoring from 0 (no movement) to 57 (normal arm function). It assesses grasp, grip, pinch, and gross arm movement.
Barthel index | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  measures a person's daily living abilities, focusing on ten areas of self-care and mobility. Scores range from 0 to 100, with higher scores denoting greater independence.
Wolf Motor Function Test | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  assess upper extremity function in individuals with neurological impairments, using 17 tasks divided into sections of time, functional ability, and strength. Scoring is on a 6-point ordinal scale, ranging from 0 ("Does not attempt with upper extremity being tested," indicating severe impairment) to 5 ("Movement appears to be normal," suggesting full functionality). Lower scores indicate greater impairment.
ultrasound assessment | pre-treatment; 1, 4, 12, and 24 weeks post-treatment
  used strain elastography to assess elasticity of shoulder muscles

CONTACTS AND LOCATIONS:
Overall Officials: Shu-mei Yang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Physical Medicine & Rehabilitation , National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Haghighat S, Khosravi M, Saadatnia M, Hashemijaazi M. Effect of Extracorporeal Shockwave Therapy on Pain Management of Patients with Post-Stroke Hemiplegic Shoulder Pain: A Prospective Randomized Controlled Trial. Adv Biomed Res. 2023 Aug 31;12:216. doi: 10.4103/abr.abr_279_21. eCollection 2023. PMID 38073721
- [Background] Wu YT, Chang CN, Chen YM, Hu GC. Comparison of the effect of focused and radial extracorporeal shock waves on spastic equinus in patients with stroke: a randomized controlled trial. Eur J Phys Rehabil Med. 2018 Aug;54(4):518-525. doi: 10.23736/S1973-9087.17.04801-8. Epub 2017 Oct 25. PMID 29072044
- [Background] Yoon SH, Shin MK, Choi EJ, Kang HJ. Effective Site for the Application of Extracorporeal Shock-Wave Therapy on Spasticity in Chronic Stroke: Muscle Belly or Myotendinous Junction. Ann Rehabil Med. 2017 Aug;41(4):547-555. doi: 10.5535/arm.2017.41.4.547. Epub 2017 Aug 31. PMID 28971038
- [Background] Li G, Yuan W, Liu G, Qiao L, Zhang Y, Wang Y, Wang W, Zhao M, Wang Y, Wang J. Effects of radial extracorporeal shockwave therapy on spasticity of upper-limb agonist/antagonist muscles in patients affected by stroke: a randomized, single-blind clinical trial. Age Ageing. 2020 Feb 27;49(2):246-252. doi: 10.1093/ageing/afz159. PMID 31846499